CLINICAL TRIAL: NCT01941758
Title: A Pilot Single Arm Study of High-Dose Influenza Vaccine Immunogenicity in Patients With Central Nervous System Tumors
Brief Title: High-Dose Trivalent Influenza Vaccine in Inducing Immune Response Patients With Central Nervous System Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00024870; NCI-2013-01740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97413 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Basic science (trivalent influenza vaccine) (Experimental): Patients receive trivalent influenza vaccine on day 1.
  Interventions: Biological: trivalent influenza vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trivalent influenza vaccine
  Other Names: Flushield; Fluvirin; Fluzone; Influenza Vaccine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies high-dose trivalent influenza vaccine in inducing immune response patients with central nervous system tumors. Studying samples of blood in the laboratory from patients receiving trivalent influenza vaccine may help doctors learn more about the effects of trivalent influenza vaccine on cells. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the immunogenicity of high-dose influenza vaccination in patients with central nervous system tumors.

SECONDARY OBJECTIVES:

I. To assess the geometric mean titer (GMT) in patients after administration of high-dose influenza vaccination compared to previously determined geometric mean titer (GMT) among 38 patients receiving the standard yearly influenza vaccination.

II. To assess the seroconversion rates (i.e. four-fold rise in titer) compared to previously determined seroconversion following administration of the standard yearly influenza vaccination.

III. To assess the seroprotection rates (i.e. post-vaccination titer >= 1:40) compared to previously determined seroconversion and seroprotection following administration of the standard yearly influenza vaccination.

TERTIARY OBJECTIVES:

I. To assess the relationship between serologic markers of immune function and response to high-dose vaccination.

OUTLINE:

Patients receive trivalent influenza vaccine on day 1.

After completion of study, patients are followed up at 28 days and/or 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of a primary central nervous system tumor
* Patients must be eligible to receive the influenza vaccine
* Patients must be willing to receive the Fluzone® high-dose seasonal influenza vaccine
* Patients must be willing and able to sign an Institutional Review Board (IRB)-approved written informed consent document

Exclusion Criteria:

* Patients unable to receive the high-dose influenza vaccine due to history of allergy to egg proteins, allergy to influenza vaccine component, acute febrile illness at the time of proposed vaccine administration, history of clinically or virologically confirmed influenza infection in the previous 6 months, contraindication to intramuscular injections, Guillain-Barré syndrome, or other contraindication to the vaccine
* Patients who have received the 2013-2014 annual influenza vaccine prior to being considered for enrollment on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Estimation of geometric mean titer (GMT) seroconversion, defined as the percentage of patients with at least a four-fold increase in hemagglutinin inhibition (HI) antibodies | Baseline
Estimation of GMT seroconversion, defined as the percentage of patients with at least a four-fold increase in HI antibodies | Day 28

SECONDARY OUTCOMES:
GMT | Up to 3 months
  Continuous values will be analyzed using Wilcoxon rank sum tests to compare high dose influenza vaccine to previously reported data on immunogenicity to the standard trivalent inactivated vaccine.
Seroconversion | Up to 3 months
  Categorical variables will be analyzed using chi-square or Fisher exact tests when necessary or appropriate.
Seroprotection rate, defined as the percentage of patients with a serum HI antibody of at least 1:40 | Up to 3 months
  Categorical variables will be analyzed using chi-square or Fisher exact tests when necessary or appropriate.

OTHER OUTCOMES:
Clinical factors such as treatment, disease status, and use of glucocorticoids | Up to 3 months
  Logistic regression models adjusting for age and gender will be used to assess the relationship between seroconversion and clinical factors.
Serologic markers of immune function | Up to 3 months
  To assess the relationship between serologic markers of immune function and response to vaccination, student's t-test will be used.
Response to vaccination | Up to 3 months
  To assess the relationship between serologic markers of immune function and response to vaccination, student's t-test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina